CLINICAL TRIAL: NCT02132858
Title: Assessing Intratumoral Heterogeneity and Chemoradiation Response in Locally Advanced Rectal Cancer Utilizing Sequencing and PET/CT
Brief Title: Genetic Mutations in Blood and Tissue Samples in Predicting Response to Treatment in Patients With Locally Advanced Rectal Cancer Undergoing Chemoradiation
Status: Completed | Type: Observational
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CGI-066; NCI-2014-00719 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CGI-066 (Other: Fox Chase Cancer Center); P30CA006927 (NIH)
Record Dates: First submitted 2014-05-06; First posted 2014-05-07 (Estimated); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Mucinous Adenocarcinoma of the Rectum; Recurrent Rectal Cancer; Signet Ring Adenocarcinoma of the Rectum; Stage IIA Rectal Cancer; Stage IIB Rectal Cancer; Stage IIC Rectal Cancer; Stage IIIA Rectal Cancer; Stage IIIB Rectal Cancer; Stage IIIC Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ancillary-Correlative (genetic mutation analysis): Patients undergo collection of blood and tissue samples for analysis via sequencing.
  Interventions: Other: cytology specimen collection procedure; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: cytology specimen collection procedure — Correlative studies
  Other Names: cytologic sampling
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies genetic mutations in blood and tissue samples to see if they can be used to predict treatment response in patients with locally advanced rectal cancer undergoing chemoradiation. Studying samples of blood and tumor tissue in the laboratory from patients with cancer may help doctors learn more about genetic mutations or changes that occur in deoxyribonucleic acid (DNA) and help doctors understand how patients respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the tumor-specific mutation(s) detected using the CancerCode™ mutation panel as a predictor of pathologic response to chemoradiation for patients with rectal adenocarcinoma undergoing chemoradiation.

SECONDARY OBJECTIVES:

I. To assess the feasibility of utilizing biopsy specimens from locally advanced rectal adenocarcinoma to perform CancerCode™ mutation panel genetic testing.

II. To assess disease-free survival (DFS) and overall survival (OS) of patients treated on study.

III. To collect pilot data regarding the clonal heterogeneity of rectal adenocarcinoma, and the relationship of this heterogeneity with treatment response.

IV. To evaluate the treatment response utilizing multiple fludeoxyglucose F 18-positron emission tomography (FDG-PET) parameters including heterogeneity and textural features as an exploratory study.

OUTLINE:

Patients undergo collection of blood and tissue samples for analysis via sequencing.

After completion of study, patients are followed up every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced rectal adenocarcinoma: T3-4NanyM0 or TanyN1-2M0
* Radiologically measurable or clinically evaluable disease
* Provide informed written consent
* Willing to return to enrolling medical site for all study assessments

Exclusion Criteria:

* Chemotherapy within 5 years prior to registration; (hormonal therapy is allowable if the disease free interval is >= 5 years)
* Any prior pelvic radiation
* Patients who are at high risk of complications from temporarily discontinuing anticoagulation for rectal cancer biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-07; Primary Completion 2022-04-08 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Proportion of the randomly chosen samples that are successfully sequenced | Up to 3 years
  If >= 90% of the specimens (at least 72 out of 80) are useable, the method will be considered feasible.
Tumor response measured using the tumor regression grading system | Up to 3 years
  Whether mutations in any gene on the CancerCode mutation panel are associated with tumor response will be assessed. In each sample, the presence or absence of mutations (0/1) for each gene on the panel will be evaluated. Each gene will be tested separately for its association with tumor response using a two-sample Mann-Whitney-Wilcoxon test with a type-I error of 0.05 for a two-sided test.

SECONDARY OUTCOMES:
Tumor heterogeneity in patients with partial response to radiation | Up to 3 years
  Whether there are differences in the mutation profiles in the 4 tumor samples will be assessed, with differences being considered evidence of possible heterogeneity.

OTHER OUTCOMES:
Progression-free survival (PFS) | Up to 3 years
  PFS will be calculated using the methods of Kaplan and Meier. If promising mutations are identified, survival between mutation positive and negative patients will be compared using the log-rank test.
Overall survival | Up to 3 years
  OS will be calculated using the methods of Kaplan and Meier. If promising mutations are identified, survival between mutation positive and negative patients will be compared using the log-rank test.
Changes in mutation profiles | Baseline to up to 3 years
  Any differences between pre- and post- test results (a different mutation status for any gene on the panel) will be considered evidence of a change. The overall proportion of patients exhibiting pre-post differences will be characterized, and particular genes of interest may be tested individually with an exact test of marginal homogeneity.
PET-computed tomography parameters | Up to 3 years
  Maximum standardized uptake value will be calculated, as well as textural measures such as coarseness, busyness, contrast, and complexity. The Mann-Whitney-Wilcoxon tests will be used to examine association between image measures and response. Image measures before and after radiation using the Wilcoxon signed rank test for paired data will be compared and differences in textural measures across tumor grades 0-3 will be assessed using the Kruskal-Wallis test. Associations between textural measures and tumor mutation profiles will be explored, also using non-parametric tests.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Meyer, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States